CLINICAL TRIAL: NCT00827892
Title: Safety of Pioglitazone for Hematoma Resolution In Intracerebral Hemorrhage
Acronym: SHRINC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Nicole Gonzales, Assistant Professor - Neurology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-08-0410; P50 NS044227-5; P50NS044227 (NIH)
Record Dates: First submitted 2009-01-21; First posted 2009-01-23 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral Hemorrhage; Treatment; MRI
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Pioglitazone
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Drug: Pioglitazone — Escalating doses for 3 days, then 30 mg orally daily for the duration of the study as determined by MRI
  Other Names: Actos
  Arms: 1
Drug: Placebo Control — Lactose Capsule administered by mouth daily for the duration of the study as determined by MRI
  Arms: 2

SUMMARY:
Intracerebral hemorrhage (ICH) is a devastating disease with less than 20% of survivors being independent at 6 months. There is currently no approved treatment for ICH which has been shown to improve outcomes. In an effort to develop a new treatment for ICH, this research focuses on a different aspect of ICH treatment which has not yet been evaluated: enhancing absorption of the blood clot with medication.

DETAILED DESCRIPTION:
Intracerebral hemorrhage (ICH) remains a devastating disease and current treatment options lag far behind those for ischemic stroke. Current treatment efforts for ICH are targeted towards the primary brain injury caused by the hemorrhage and growth of the hematoma. This research targets the secondary injury caused by the persistence of toxic blood degradation products in the brain parenchyma.

Based on preclinical work in our lab, the peroxisome proliferator activated receptor-gamma (PPARγ), a member of the nuclear receptor superfamily, represents a possible target for the treatment of ICH aimed at promoting hematoma absorption, limiting the pro-inflammatory response, and protecting salvageable tissue from the damage produced by the persistence of toxic blood degradation products.

Our primary specific aim is to assess the safety of the PPARγ agonist, pioglitazone (PIO) in increasing doses for 3 days, when administered to patients with ICH within 24 hrs of symptom onset. Secondarily, we aim to determine the duration of treatment of PIO for hematoma/edema resolution in ICH. Lastly, we aim to determine whether speed of hematoma/edema resolution in ICH represents a radiographic biological marker of activity which can be correlated with clinical outcome and treatment effect of PIO. The ultimate purpose is to provide baseline data on an aspect of ICH which has not been previously targeted for treatment in an effort to develop a safe and effective treatment strategy that may be practical and applicable for both specialized stroke centers and community hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-80 years
2. clinical presentation of spontaneous ICH
3. CT scan compatible with spontaneous ICH
4. Time to PIO treatment ≤ 24 hours from symptom onset
5. GCS ≥ 6 on initial presentation OR improvement to a GCS ≥ 6 within the time frame for enrollment
6. Hematoma volume ≥ 5cc on initial head CT.

Exclusion Criteria:

1. Participation in another investigational trial in the previous 30 days
2. Patient will undergo surgical evacuation of ICH (ventriculostomy does NOT exclude patient)
3. Inability to undergo neuroimaging with MRI (e.g. pacer, recent stent, inability to lie flat)

   a. If patient has mild claustrophobia or agitation amenable to mild sedation (1-2mg lorazepam IV or 5-10mg diazepam PO), he or she may be considered for enrollment. If, however, the patient has severe claustrophobia or agitation, he or she should not be considered for enrollment.
4. GCS < 6
5. Baseline mRS ≥ 3
6. Primary intraventricular hemorrhage
7. ICH due to coagulopathy (PT > 15 sec or INR > 1.3, PTT > 36) or trauma
8. History of intolerance or allergy to any TZD
9. Thrombocytopenia: platelet count < 100,000
10. Clinically significant hepatic disease as demonstrated by history, clinical exam (ascites, varices), or laboratory findings (LFTs ≥ 2x normal, coagulopathy as described above)
11. Co-morbid conditions, which in the opinion of the investigator, are likely to complicate therapy including but not limited to:

    1. A history of NYHA class II, III, or IV CHF
    2. clinically significant arrhythmia
    3. end stage AIDS
12. Pregnancy as determined by a urine pregnancy test
13. Severe anemia at presentation: hemoglobin < 10 g/dL or hematocrit < 30%
14. Malignancy (history of or active)
15. Patient unlikely, in the investigator's opinion, to complete the study and return for follow-up visits for any reason

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-03; Primary Completion 2013-04 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The primary measure of safety will be mortality at discharge. | At hospital discharge or Day 14, whichever occurs first.

SECONDARY OUTCOMES:
Secondary measures of safety will include mortality at 3 months and 6 months, symptomatic cerebral edema during hospitalization, clinically significant congestive heart failure, edema, hypoglycemia, anemia, and hepatotoxicity. | 3 months, 6 months, and during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Nicole R Gonzales, MD, Principal Investigator — University of Texas Medical School-Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Zhao X, Sun G, Zhang J, Strong R, Song W, Gonzales N, Grotta JC, Aronowski J. Hematoma resolution as a target for intracerebral hemorrhage treatment: role for peroxisome proliferator-activated receptor gamma in microglia/macrophages. Ann Neurol. 2007 Apr;61(4):352-62. doi: 10.1002/ana.21097. PMID 17457822
- [Background] Zhao X, Grotta J, Gonzales N, Aronowski J. Hematoma resolution as a therapeutic target: the role of microglia/macrophages. Stroke. 2009 Mar;40(3 Suppl):S92-4. doi: 10.1161/STROKEAHA.108.533158. Epub 2008 Dec 8. PMID 19064796